CLINICAL TRIAL: NCT02741687
Title: Prevention of Stress Hyperglycemia With the Use of DPP-4 Inhibitors in Non-diabetic Patients Undergoing Non-cardiac Surgery, a Pilot Study
Brief Title: Sitagliptin in Non-Diabetic Patients Undergoing General Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Maya Fayfman, Instructor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00087357
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Hyperglycemia
Keywords: stress hyperglycemia; blood glucose
MeSH Terms: conditions — Hyperglycemia | interventions — Sitagliptin Phosphate; Insulin Lispro; Insulin Aspart; Insulin Detemir; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin Arm (Experimental): Participants will receive sitagliptin beginning the day prior to surgery and continuing daily during hospitalization (up to 10 days post-surgery).
  Point of care (POC) testing will be done four times daily, before meals and at bedtime, or every 6 hours for patients who are not eating (NPO). Patients developing hyperglycemia during or after surgery will be treated with insulin per standard of care.
  Patients with fasting and/or premeal blood glucose levels >180 mg/dl will receive supplemental insulin provided on a sliding scale. Patients with two consecutive fasting and/or premeal blood glucose levels >180 mg/dl, or with average daily blood glucose levels >180 mg/dl will be started on rescue therapy with subcutaneous insulin once daily plus correction doses by a sliding scale.
  Interventions: Drug: Sitagliptin; Drug: Supplemental insulin (insulin lispro); Drug: Supplemental insulin (insulin aspart); Drug: Long acting basal insulin (insulin detemir); Drug: Long acting basal insulin (insulin glargine)
- Placebo Arm (Placebo Comparator): Participants will receive a placebo tablet beginning the day prior to surgery and continuing daily during hospitalization (up to 10 days post-surgery).
  Point of care (POC) testing will be done four times daily, before meals and at bedtime, or every 6 hours for patients who are not eating (NPO). Patients developing hyperglycemia during or after surgery will be treated with insulin per standard of care.
  Patients with fasting and/or premeal blood glucose levels >180 mg/dl will receive supplemental insulin provided on a sliding scale. Patients with two consecutive fasting and/or premeal blood glucose levels >180 mg/dl, or with average daily blood glucose levels >180 mg/dl will be started on rescue therapy with subcutaneous insulin once daily plus correction doses by a sliding scale.
  Interventions: Drug: Placebo; Drug: Supplemental insulin (insulin lispro); Drug: Supplemental insulin (insulin aspart); Drug: Long acting basal insulin (insulin detemir); Drug: Long acting basal insulin (insulin glargine)

INTERVENTIONS:
Drug: Sitagliptin — Participants will take 100 mg/day for patients with glomerular filtration rate (GFR) > 50 and 50 mg/day for GFR 30 - 49, beginning on the day prior to surgery and continuing through hospitalization, up to 10 days.
  Other Names: Januvia
  Arms: Sitagliptin Arm
Drug: Placebo — Participants will take one pill daily beginning on the day prior to surgery and continuing through hospitalization, up to 10 days.
  Arms: Placebo Arm
Drug: Supplemental insulin (insulin lispro) — Supplemental insulin lispro will be administered before meals, in addition to scheduled insulin dose, following the supplemental insulin scale protocol. At bedtime, half of supplemental sliding scale insulin starting at blood glucose (BG) >240 mg/dL will be given. If a patient is unable to eat, supplemental insulin will be administered every 6 hours with the lowest number of units for that appropriate BG level.
  For subjects receiving supplemental insulin lispro with BG levels greater than 180 mg/dL, the supplemental insulin scale is as follows:
  * BG between 181-220 mg/dL; 2-4 units of insulin lispro
  * BG between 221-260 mg/dL; 3-5 units of insulin lispro
  * BG between 261-300 mg/dL; 4-6 units of insulin lispro
  * BG between 301-350 mg/dL; 5-7 units of insulin lispro
  * BG between 351-400 mg/dL; 6-8 units of insulin lispro
  * BG > 400 mg/dL; 7-9 units of insulin lispro
  Other Names: Humalog
Drug: Supplemental insulin (insulin aspart) — Supplemental insulin aspart will be administered before meals, in addition to scheduled insulin dose, following the supplemental insulin scale protocol. At bedtime, half of supplemental sliding scale insulin starting at blood glucose (BG) >240 mg/dL will be given. If a patient is unable to eat, supplemental insulin will be administered every 6 hours with the lowest number of units for that appropriate BG level.
  For subjects receiving supplemental insulin aspart with BG levels greater than 180 mg/dL, the supplemental insulin scale is as follows:
  * BG between 181-220 mg/dL; 2-4 units of insulin lispro
  * BG between 221-260 mg/dL; 3-5 units of insulin lispro
  * BG between 261-300 mg/dL; 4-6 units of insulin lispro
  * BG between 301-350 mg/dL; 5-7 units of insulin lispro
  * BG between 351-400 mg/dL; 6-8 units of insulin lispro
  * BG > 400 mg/dL; 7-9 units of insulin lispro
  Other Names: NovoLog
Drug: Long acting basal insulin (insulin detemir) — Long acting basal insulin therapy will be provided as needed, and will be given once daily, at the same time of day. Participants with blood glucose (BG) >180 mg/dL= start detemir at 0.2 units per kg weight per day and will follow the following adjustment schedule:
  * Fasting and pre-meal BG between 100-180 mg/dl without hypoglycemia the previous day: no change
  * Fasting and pre-meal BG between >180-240 mg/dl: increase detemir or glargine dose by 10% every day
  * Fasting and pre-meal BG >241 mg/dl: increase detemir or glargine dose by 20% every day
  * Fasting and pre-meal BG <100 mg/dl: reduce detemir or glargine by 20% or stop if patient is already on less than 0.1 units/kg of body weight
  Other Names: Levemir
Drug: Long acting basal insulin (insulin glargine) — Long acting basal insulin therapy will be provided as needed, and will be given once daily, at the same time of day. Participants with blood glucose (BG) >180 mg/dL= start detemir at 0.2 units per kg weight per day and will follow the following adjustment schedule:
  * Fasting and pre-meal BG between 100-180 mg/dl without hypoglycemia the previous day: no change
  * Fasting and pre-meal BG between >180-240 mg/dl: increase detemir or glargine dose by 10% every day
  * Fasting and pre-meal BG >241 mg/dl: increase detemir or glargine dose by 20% every day
  * Fasting and pre-meal BG <100 mg/dl: reduce detemir or glargine by 20% or stop if patient is already on less than 0.1 units/kg of body weight
  Other Names: Lantus

SUMMARY:
The purpose of this study is to compare sitagliptin with a placebo for the prevention of high glucose after general surgery.

DETAILED DESCRIPTION:
Approximately 30-40% of hospitalized patients will develop stress hyperglycemia (high glucose in response to surgery or illness). High glucose is linked to an increased risk of hospital complications including wound infection, kidney failure and death. Patients with high glucose are treated with insulin given through an arm vein or by frequent insulin injections under the skin. Recent studies have found that inpatient therapy with oral dipeptidyl peptidase-4 inhibitor (DPP4-I) is an effective alternative to insulin in improving glycemic control with low risk of hypoglycemia in general medicine and surgical patients.

Sitagliptin is an oral medication approved by the Food and Drug Administration (FDA) to treat patients with diabetes. The aim of this study is to determine whether treatment with sitagliptin once daily can prevent the development of stress hyperglycemia during the postoperative period in non-diabetic patients undergoing general surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing non-cardiac surgery
* No previous history of diabetes or hyperglycemia
* Fasting blood glucose level of <126 mg/dl
* Blood glucose <126mg/dl at the time of randomization (could occur at any time of the day)

Exclusion Criteria:

* History of hyperglycemia (blood glucose equal to or above 126 mg/dl or HbA1C greater than 6.5%) or previous treatment with oral antidiabetic agents or insulin
* Patients undergoing cardiac surgery
* Patients anticipated to require ICU care following surgery
* Severely impaired renal function (GFR < 30 ml/min) or clinically significant hepatic failure
* Moribund patients and those at imminent risk of death (brain death or cardiac standstill)
* Patients with gastrointestinal obstruction or adynamic ileus or those expected to require gastrointestinal suction
* Patients with clinically relevant pancreatic or gallbladder disease
* Treatment with oral (> 5 mg/day) or injectable corticosteroid
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Pregnancy or breast-feeding at time of enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maya Fayfman, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital and Grady Hospital in Atlanta, Georgia between June 2016 and March 2017.
Pre-assignment Details: A total of 97 patients consented to be in the study and one participant withdrew prior to randomization. After subsequent failure to meet eligibility criteria (such as surgery being cancelled or postponed) and voluntary participant withdrawals prior to receiving the study medication there were 80 participants who received the study intervention.
Groups:
- Placebo: Participants received a placebo identical to sitagliptin beginning on the day before surgery and continuing daily during hospitalization (up to 10 days post surgery)
- Sitagliptin: Participants received sitagliptin beginning on the day before surgery and continuing daily during hospitalization (up to 10 days post surgery)
Period: Overall Study
Arm/Group | Placebo | Sitagliptin
Started | 36 | 44
Completed | 36 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who began the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sitagliptin | Total
Number analyzed (Participants) | 36 | 44 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (14.5) | 51.1 (12.8) | 48.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 18 | 25 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 26 | 32 | 58
  Race: White | 8 | 11 | 19
  Race: Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 44 | 80
Surgery type [Count of Participants; unit: Participants]
  Orthopedic | 6 | 11 | 17
  Genitourinary | 9 | 14 | 23
  Gastrointestinal | 3 | 3 | 6
  Neurologic | 4 | 5 | 9
  Oral maxillofacial surgery | 4 | 1 | 5
  Thoracic | 2 | 2 | 4
  Burn/Wound | 1 | 4 | 5
  Vascular | 0 | 1 | 1
  gynecologic | 7 | 3 | 10
ASA Status [Count of Participants; unit: Participants] — The American Society of Anesthesiology (ASA) Physical Status Classification is a method of assessing patients prior to surgery. The following categories are used:
  1. = Healthy person
  2. = Mild systemic disease
  3. = Severe systemic disease
  4. = Severe systemic disease that is a constant threat to life
  5. = A moribund person who is not expected to survive with the operation
  6. = A declared brain-dead person whose organs are being removed for donor purposes
  Participants
    ASA status = 1 | 4 | 4 | 8
    ASA status = 2 | 17 | 22 | 39
    ASA status = 3 | 9 | 13 | 22
    Unknown | 6 | 5 | 11
Admission blood glucose [Mean (Standard Deviation); unit: mg/dl] | 98.5 (20.0) | 107.6 (25.3) | 103.6 (23.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Stress Hyperglycemia
Description: The number of participants with at least one episode of stress hyperglycemia. Stress hyperglycemia is defined as a blood glucose > 180 mg/dL.
Time Frame: Up to time of discharge from hospital, an average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 36 | 44
Participants | 7 | 5

2. Secondary Outcome: Number of Patients Requiring Supplemental, Subcutaneous Insulin
Description: Number of patients requiring subcutaneous insulin, either sliding scale insulin or basal insulin
Time Frame: Up to time of discharge from hospital, an average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 36 | 44
Participants | 0 | 1

3. Secondary Outcome: Total Daily Dose of Insulin for Patients Requiring Supplemental Insulin
Description: Total daily dose of insulin for patients requiring supplemental insulin during surgery and recovery in participants receiving sitagliptin and those receiving the placebo
Time Frame: Up to time of discharge from hospital, an average of 10 days
Population: The population for this analysis is limited to participants who received insulin during their hospital stay following surgery.
Measure: Number; unit: international units of insulin
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 0 | 1
international units of insulin |  | 5

4. Secondary Outcome: Length of Hospital Stay
Description: Total length of hospital stay
Time Frame: Up to time of discharge from hospital, an average of 10 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 36 | 44
days | 9 [5 to 12] | 11 [7 to 14]

5. Secondary Outcome: Number of Participants With Hypoglycemic Events
Description: Number of participants experiencing at least one episode of mild hypoglycemia (blood glucose < 70 mg/dL) or clinically significant hypoglycemia (blood glucose < 54 mg/dL)
Time Frame: Up to time of discharge from hospital, an average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 36 | 44
Participants
  Mild hypoglycemia | 2 | 5
  Clinically significant hypoglycemia | 0 | 0

6. Secondary Outcome: Number of Patients Transferred to the ICU Immediately After Surgery or During Hospitalization
Description: The number of patients who were transferred to the ICU immediately following surgery or anytime while hospitalized after surgery.
Time Frame: Up to time of discharge from hospital, an average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 36 | 44
Participants | 1 | 2

7. Secondary Outcome: Number of Days in the ICU
Description: The number of days a participant spent in the ICU following surgery, when transfer to the ICU was required.
Time Frame: Up to time of discharge from hospital, an average of 10 days
Population: This analysis includes participants who were transferred to the ICU following surgery.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 1 | 2
days | 2.0 [2.0 to 2.0] | 1.5 [1.0 to 2.0]

8. Secondary Outcome: Number of Participants With Hospital Readmissions After Discharge
Description: Readmissions to the study hospital occurring within 30 days of hospital discharge were documented. There were no follow up phone calls or appointments with participants so any hospital readmissions to hospitals other than the one where the surgery occurred are not known.
Time Frame: Up to 40 days (average time of discharge from the hospital plus 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 36 | 44
Participants | 0 | 1

9. Secondary Outcome: Number of Participants With Emergency Room Visits After Discharge
Description: Emergency room visits to the study hospital occurring within 30 days of hospital discharge were documented. There were no follow up phone calls or appointments with participants so any emergency room visits to hospitals other than the one where the surgery occurred are not known.
Time Frame: Up to 40 days (average time of discharge from the hospital plus 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 36 | 44
Participants | 0 | 0

10. Secondary Outcome: Number of Participants Experiencing Complications
Description: The number of subjects who experience complications including: wound infection, respiratory failure, pneumonia, acute kidney injury with a rise in creatinine by 38 micromoles/Liter from baseline, major adverse cardiac events, bacterial septic infection, and death. Participants will be followed for 30 days following hospital discharge and all complications will be documented.
Time Frame: Up to 40 days (average time of discharge from the hospital plus 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 36 | 44
Participants
  Wound infection | 0 | 0
  Respiratory failure | 0 | 0
  Pneumonia | 0 | 0
  Acute kidney injury | 1 | 1
  Cardiac event | 0 | 0
  Bacterial septic infection | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the time a participants gave informed consent through 30 days after discharge from the hospital.
Arm/Group | Placebo | Sitagliptin
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/44
Other Adverse Events (participants affected / at risk) | 5/36 | 8/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Sitagliptin (N=44)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Due to anesthesia medication
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Sitagliptin (N=44)
Ileus (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1
Chest pain (Cardiac disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Repeat operation (Surgical and medical procedures) | 1 | 2
Tachycardia with anemia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT02741687/Prot_SAP_000.pdf